CLINICAL TRIAL: NCT04046146
Title: Near InfraRed Fluorescence Using Indocyanine Green and Magnetic Resonance Lymphography of Lymphatic Transport
Acronym: NIR-ICG MRL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Homaira Rahimi, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY3891
Record Dates: First submitted 2019-07-23; First posted 2019-08-06 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Healthy Volunteers; Lymphatic Transport; Imaging; Indocyanine Green; Gadolinium; ICG; GAD; NIR-ICG; rhuematoid arthritis; NIR
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NIR-ICG MRL (Experimental): We may ask healthy subjects to return for up to four injection sessions for the study. The first injection session will consist of intradermal injection of ICG into the webspaces of the hand as done in our previous studies followed by NIR camera imaging. The second session will consist of intradermal gadolinium injection and intravenous (IV) iron contrast agent followed by MRI imaging approximately 1 week after the first session. The third session will occur at minimum eight weeks later and entail intra-articular ICG injection in order to evaluate drainage via the lymphatics. The MCP joints will be identified in the non-dominant hand and injected with ICG. Approximately one week later, the fourth session will compromise of intra-articular gadolinium injection and IV iron contrast to confirm lymphatic drainage. The MCP joints of the non-dominant hand will again be identified and injected with gadolinium.
  Interventions: Drug: Indocyanine Green; Device: MultiSpectral Imaging System

INTERVENTIONS:
Drug: Indocyanine Green — A trained physician will inject 0.1 ml of Indocyanine Green into the web spaces of the hands in both upper extremities. Subjects may have up to five study visits to confirm feasibility, safety, and reproducibility.
  Other Names: ICG; IC-Green; 17478-701-02
Device: MultiSpectral Imaging System — Once the Indocyanine Green is injected, the contrast is expected to fluoresce underneath the MultiSpectral Imaging System. Multispectral video and still images will be recorded at the study visits.
  Other Names: MSImager

SUMMARY:
Lymphatic transport will be examined using Near InfraRed Indocyanine Green fluorescence imaging (NIR-ICG) and magnetic resonance lymphography (MRL) of the upper extremities. The purpose of the study is to establish if NIR-ICG is a valid clinical outcome for quantifying lymphatic vessel drainage.

DETAILED DESCRIPTION:
Lymphedema from various etiologies (i.e. infection, cancer, surgery, and rheumatoid arthritis) remains a major health concern. Efforts to develop effective treatments for this condition have been limited by the absence of quantitative outcome measures for lymphatic function. Published articles have supported the fact that human lymphatic contractions can be readily visualized after intradermal administration of micrograms of Indocyanine Green using laser-induced fluorescence. We recently demonstrated the feasibility of NIR imaging to quantify lymphatic drainage in the hands, wrists and forearms of healthy volunteers following intradermal web space ICG injection into the hand . To establish this emerging technology as a valid clinical outcome measure, however, we must address two major questions that confound interpretation of the imaging results: 1) are the ICG filled vessels lymphatic vessels and/or small veins?; and 2) does NIR-ICG imaging following web space injection fully capture lymphatic flow from the metacarpophalangeal (MCP) joints that are most commonly involved in RA? To answer these questions, healthy patients will be recruited to have intradermal and intra-articular injections of ICG and gadolinium followed by an imaging sessions (NIR or magnetic resonance imaging) to measure lymphatic contraction rates and flow.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent.
* Subjects must be 18 years old or older.

Exclusion Criteria:

* Active systemic disorders or inflammatory conditions (i.e., chronic infections with hepatitis B, hepatitis C or HIV) that would confound the study results.
* Known sensitivity to iodine because of residual iodide in indocyanine green
* Known sensitivity to gadolinium
* Any history of kidney disease
* Pregnant women should not participate; pregnancy tests will not be performed.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Manual lymphatic vessel counts via assessment of 2D images of NIR-ICG compared to MRI. Unit of measure: # lymphatic vessels/hand | 12 months
  Vessel location and numbers will be identified using 2D still images from the NIR scanning sessions and with 2D MR images. These images will be superimposed upon each other in order to confirm concordance of lymphatic vessels. Number of lymphatic vessels in the hands will be manually counted.
Lymphatic contraction rate measured via NIR ICG camera. Unit of measure: # contraction/minute | 12 months
  Images collected from NIR scanning sessions will be analyzed to determine lymphatic contraction rate by identifying number of contractions per minute.
ICG clearance measured from hand using NIR ICG images. Unit of measure: (% difference Visit 1 from Visit 2) | 12 months
  2D still images collected from NIR scanning sessions will be analyzed to determine ICG clearance by comparing the % difference from visit 1 to visit 2.

CONTACTS AND LOCATIONS:
Overall Officials: Homaira Rahimi, MD, MTR, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Information of any type may be shared with researchers at other institutions. Subjects will be made aware of this in the informed consent form.

REFERENCES:
- [Derived] Kenney HM, Dieudonne G, Yee S, Maki JH, Wood RW, Schwarz EM, Ritchlin CT, Rahimi H. Near-Infrared Imaging of Indocyanine Green Identifies Novel Routes of Lymphatic Drainage from Metacarpophalangeal Joints in Healthy Human Hands. Lymphat Res Biol. 2023 Aug;21(4):388-395. doi: 10.1089/lrb.2022.0026. Epub 2023 Feb 20. PMID 36809077